CLINICAL TRIAL: NCT03420196
Title: Efficacy of a Supervised Physical Therapy Rehabilitation Program vs Nonsupervised on Pain, Disability, Quality of Life and Kinesiophobia in Patients With Non-specific Low Back Pain
Brief Title: Efficacy of a Supervised Physical Therapy Rehabilitation Program vs Nonsupervised in Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-476
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain; Physical Activity
Keywords: low back pain; physical therapy; randomized clinical trial; exercise program
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Rehabilitation program (Experimental): It will be consist in a supervised exercise program by physical therapist, including the following structures: diaphragm, tranverse abdominis muscle, pelvic, gluteus, CORE and spinal mobility
  Interventions: Other: Supervised exercise program
- Nonsupervised rehabilitation program (Active Comparator): It will consist in an exercise program for home, nonsupervised, including the following structures: diaphragm, tranverse abdominis muscle, pelvic, gluteus, CORE and spinal mobility. The patients will perform an exercise program at home.
  Interventions: Other: Non supervised exercise program

INTERVENTIONS:
Other: Supervised exercise program — It will consist in a supervised exercise program, including the following exercises:
  * Diaphragmatic breathing.
  * Transverse abdomLateral leg raise for gluteus mediuminis muscle activation.
  * Pelvic swing.
  * Gluteus bridge.
  * Spinal mobility.
  * Spinal extensor muscles strengthening
  * Frontal plank
  * Side plank.
  * Lateral leg raise for gluteus medium
  Arms: Supervised Rehabilitation program
Other: Non supervised exercise program — It will consist in a non supervised exercise program, including the following exercises:
  * Diaphragmatic breathing.
  * Transverse abdomLateral leg raise for gluteus mediuminis muscle activation.
  * Pelvic swing.
  * Gluteus bridge.
  * Spinal mobility.
  * Spinal extensor muscles strengthening
  * Frontal plank
  * Side plank.
  * Lateral leg raise for gluteus medium
  Arms: Nonsupervised rehabilitation program

SUMMARY:
This study compares the efficacy of a supervised rehabilitation program vs a non supervised rehabilitation program on pain, disability, quality of life and kinesiophobia in patients with non-specific low back pain.

DETAILED DESCRIPTION:
Low back pain is one of the most common problems of population, being a priority for health systems. It has got a high prevalence and recurrence, affecting in a social and economic way, and, it is one of principal causes of laboral absenteism. A randomized clinical trial will be conducted comparing a supervised physical therapy rehabilitation program vs a non supervised rehabilitation program.

Objective: to compare the efficacy of a supervised rehabilitation program vs a non supervised rehabilitation program in patients with non-specific low back pain.

Methods: Sixt-four subjects with chronic non-specific low back pain will be assigned to supervised rehabilitation program or non supervised rehabilitation program during 4 weeks (5 sessions/week). Outcomes measures will be the following: disability, pain intensity, fear of movement, quality of life, McQuade Test, and lumbar mobility flexion.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific low back pain persisting ≥ 3 months.
* Age between 18 and 65 years.
* A score ≥ 4 in Roland Morris Disability Questionnaire.
* Not currently receiving physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis.
* Presence of clinical signs of radiculopathy.
* Diagnosis of spondylolisthesis.
* Diagnosis of fibromyalgia.
* Treatment with corticosteroid or pharmachological medication within the paset 2 weeks.
* A history of spinal surgery.
* Central or peripheral nervous system disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ) | at baseline,immediate post-treatment and at 6 months
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities

SECONDARY OUTCOMES:
Change from baseline in disability. Oswestry Low Back Pain Disability Index. | At baseline, immediate post-treatment and at 6 months
  It has 10 items associated to activities of daily living, each item has a puntuation fron 0 to 5 points
Change from baseline in pain intensity (Visual Analogue Scale). | At baseline, immediate post-treatment and at 6 months
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline, immediate post-treatment and at 6 months
  It is a 17-item questionnaire that measures the fear of movement and (re)injury
Change from baseline on Quality of Life. | At baseline, immediate post-treatment and at 6 months
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Change from Mcquade Test | at baseline, immediate post-treatment and at 6 months
  It measures the isometric endurance of trunk flexion muscles
Change from baseline in lumbar mobility flexion | at baseline, immediate post-treatment and at 6 months
  It is determined by measuring the finger-to-floor distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Andalusia, Spain

REFERENCES:
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Manchikanti L, Singh V, Falco FJ, Benyamin RM, Hirsch JA. Epidemiology of low back pain in adults. Neuromodulation. 2014 Oct;17 Suppl 2:3-10. doi: 10.1111/ner.12018. PMID 25395111
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Hu H, Zheng Y, Wang X, Chen B, Dong Y, Zhang J, Liu X, Gong D. Correlations between lumbar neuromuscular function and pain, lumbar disability in patients with nonspecific low back pain: A cross-sectional study. Medicine (Baltimore). 2017 Sep;96(36):e7991. doi: 10.1097/MD.0000000000007991. PMID 28885356
- [Background] Jubany J, Danneels L, Angulo-Barroso R. The influence of fatigue and chronic low back pain on muscle recruitment patterns following an unexpected external perturbation. BMC Musculoskelet Disord. 2017 Apr 19;18(1):161. doi: 10.1186/s12891-017-1523-3. PMID 28420353
- [Background] Marshall PWM, Schabrun S, Knox MF. Physical activity and the mediating effect of fear, depression, anxiety, and catastrophizing on pain related disability in people with chronic low back pain. PLoS One. 2017 Jul 7;12(7):e0180788. doi: 10.1371/journal.pone.0180788. eCollection 2017. PMID 28686644
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Roland M, Morris R. A study of the natural history of low-back pain. Part II: development of guidelines for trials of treatment in primary care. Spine (Phila Pa 1976). 1983 Mar;8(2):145-50. doi: 10.1097/00007632-198303000-00005. PMID 6222487
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470